CLINICAL TRIAL: NCT01601834
Title: A Double Blind (3rd Party Open) Randomized, Placebo Controlled, Crossover Dose Escalation Study To Investigate The Safety, Toleration And Pharmacokinetics Of Pf-06273340 In Healthy Volunteers
Brief Title: A First In Human Study In Healthy People To Evaluate Safety, Toleration And Time Course Of Plasma Concentration Of Single Oral Doses Of PF-06273340
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B5261001
Record Dates: First submitted 2012-04-27; First posted 2012-05-18 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: PAIN
Keywords: Phase 1; Single Dose; Pharmacokinetics; Safety; Toleration
MeSH Terms: conditions — Pain | interventions — PF-06273340

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1: Experimental intervention: PF-06273340 or placebo (Experimental): Subjects in Cohort 1 will receive single ascending doses of PF-06273340 or placebo to investigate the safety/tolerability and PK of PF-06273340. The effect of food on PK may also be investigated.
  Interventions: Drug: PF-06273340 or Placebo
- Cohort 2: Experimental intervention: PF-06273340 or placebo (Experimental): Subjects in Cohort 2 will receive single ascending doses of PF-06273340 or placebo to investigate the safety/tolerability and PK of PF-06273340. The effect of food on PK may also be investigated.
  Interventions: Drug: PF-06273340 or Placebo

INTERVENTIONS:
Drug: PF-06273340 or Placebo — PF-06273340 will be administered as an extemporaneously prepared solution for all doses. Correspondingly, placebo doses will be administered as solution.
  Arms: Cohort 1: Experimental intervention: PF-06273340 or placebo
Drug: PF-06273340 or Placebo — PF-06273340 will be administered as an extemporaneously prepared solution for all doses. Correspondingly, placebo doses will be administered as solution.
  Arms: Cohort 2: Experimental intervention: PF-06273340 or placebo

SUMMARY:
The purpose of this study in healthy people is to evaluate safety, toleration and time course of plasma concentration of single oral doses of PF-06273340. The effect of food on the Pharmacokinetic of PF-06273340 may also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects or female subjects of non-child bearing potential between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (e.g., gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* Screening supine blood pressure >= 140 mm Hg (systolic) or >= 90 mm Hg (diastolic), on a single measurement (confirmed by a single repeat, if necessary) following at least 5 minutes of rest.
* 12-lead ECG demonstrating QTc >450 msec at screening. If QTc exceeds 450 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility.
* Females of child bearing potential.
* Use of prescription or non-prescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Herbal supplements must be discontinued 28 days prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of 1 g/day. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
* Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing. History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Unwilling or unable to comply with the Lifestyle guidelines described in this protocol.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | 0,0.25,0.5,1,1.5,2,4,6,8,12,24,36,48,72 hours post-dose
Time of maximum concentration (Tmax) | 0,0.25,0.5,1,1.5,2,4,6,8,12,24,36,48,72 hours post-dose
Area under the plasma concentration time profile from time zero to the time of last quantifiable concentration (AUClast) | 0,0.25,0.5,1,1.5,2,4,6,8,12,24,36,48,72 hours post-dose
Area under the plasma concentration time profile from time zero extrapolated to inifinite time (AUCinf) | 0,0.25,0.5,1,1.5,2,4,6,8,12,24,36,48,72 hours post-dose
Area under the plasma concentration time profile from time zero to quantifiable concentration 24 h post dose (AUC24) | 0,0.25,0.5,1,1.5,2,4,6,8,12,24,36,48,72 hours post-dose
Apparent Clearance (CL/F) | 0,0.25,0.5,1,1.5,2,4,6,8,12,24,36,48,72 hours post-dose
Apparent Volume of Distribution (Vz/F) | 0,0.25,0.5,1,1.5,2,4,6,8,12,24,36,48,72 hours post-dose
t1/2 = Terminal Elimination half life | 0,0.25,0.5,1,1.5,2,4,6,8,12,24,36,48,72 hours post-dose
Urine: Ae24 (amount excreted in urine), Ae24% (%dose excreted in urine to time 24 h) and CLr (Renal Clearance) for selected doses | up to 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5261001&StudyName=A%20First%20In%20Human%20Study%20In%20Healthy%20People%20To%20Evaluate%20Safety%2C%20Toleration%20And%20Time%20Course%20Of%20Plasma%20Concentration%20Of%20Single%20Oral%20Dos